CLINICAL TRIAL: NCT00704964
Title: Impact of Patient Support From Medical Staff on the Adherence to Therapy With PegIntron Plus Rebetol
Brief Title: Impact of Patient Support by the Medical Staff on Adherence to Therapy With PegIntron Plus Rebetol (Study P04413)
Acronym: @dhere
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: P04413
Record Dates: First submitted 2008-06-23; First posted 2008-06-25 (Estimated); Results first posted 2011-04-21 (Estimated); Last update posted 2015-10-06 (Estimated); Status verified 2015-10

CONDITIONS: Hepatitis C; Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C; Hepatitis C, Chronic | interventions — peginterferon alfa-2b; Ribavirin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All participants: Each site will be evaluated by a site questionnaire and assigned as either a high or low participant management site. Participants are not randomized to a group. However, treatment completion rates will be evaluated based on the high vs low participant management sites.
  Interventions: Biological: PegIntron; Drug: Rebetol

INTERVENTIONS:
Biological: PegIntron — PegIntron (peginterferon alfa-2b) pen administered at a dose and frequency in accordance with approved labeling in Germany
  Other Names: PegIntron pen; peginterferon alfa-2b; SCH 54031
Drug: Rebetol — Rebetol (ribavirin) administered at a dose and frequency in accordance with approved labeling in Germany
  Other Names: ribavirin; SCH 18908

SUMMARY:
The objective of this study is to assess the impact of participant care and support on treatment adherence. PegIntron pen and Rebetol will be administered to participants with Hepatitis C Virus (HCV) in accordance with approved labeling. Sites will be categorized as providing high vs low level of participant management based on information about the level of participant support and management captured on the site questionnaire. Data on each participant will be collected by a physician on an electronic participant case report form (CRF) and by the participant via a questionnaire. Treatment completion rates will be analyzed based on the high vs low level of participant management.

The hypothesis is that Physicians investing more time and effort into participant management achieve higher treatment completion rates among their hepatitis C patients than physicians offering less participant management measures.

ELIGIBILITY:
Inclusion Criteria:

* Participants with chronic hepatitis C.

Those participating in patient assistance programs during therapy for hepatitis C.

Exclusion Criteria:

* Participants who have previously been treatment for hepatitis C (non-naïve)

Other exclusion criteria as described in local Summary of Product Characteristics (SPC).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with chronic hepatitis C treated in 44 non-university centers in Germany.
Sampling Method: Non-Probability Sample
Enrollment: 746 (Actual)
Dates: Start 2005-05; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: Each site will be evaluated by a site questionnaire and assigned as either a high or low participant management site. Participants are not randomized to a group. However, treatment completion rates will be evaluated based on the high vs low participant management sites.
  Completers are considered those with documentation who finished the study on time.
Period: Overall Study
Arm/Group | All Participants
Started | 746 (Number of participants who took at least one dose of study medication.)
Completed | 418 (Number of participants who completed therapy as scheduled.)
Not Completed | 328
Not completed — Not completed on time | 328

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 746
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.3 (11.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 297
  Male | 449
Region of Enrollment [Number; unit: participants]
  Germany | 746

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Biometrical Adherence to Therapy
Description: Adherence was defined as participants receiving at least 80% of the planned PegIntron doses, or at least 80% of the planned Rebetol doses, or participants concluding at least 80% of the planned duration of their treatment, or all three conditions.
Time Frame: Up to 48 weeks for Hepatitis C Virus (HCV) genotype 1 or 4 participants and up to 24 weeks for HCV genotype 2 or 3
Measure: Number; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 746
Participants
  PegIntron + Rebetol | 406
  PegIntron | 415
  Rebetol | 413

2. Primary Outcome: Number of Participants With Adherence to Therapy According to Physician Approximation
Description: Adherence was based on physiciant's clinical judgment.
Time Frame: Up to 48 weeks for HCV genotype 1 or 4 participants and up to 24 weeks for HCV genotype 2 or 3
Measure: Number; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 746
Participants
  PegIntron | 615
  Rebetol | 604

ADVERSE EVENTS:
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 27/746
Other Adverse Events (participants affected / at risk) | 332/746
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=746)
ANAEMIA (Blood and lymphatic system disorders) | 1 (2)
LEUKOPENIA (Blood and lymphatic system disorders) | 2 (2)
ACUTE CORONARY SYNDROME (Cardiac disorders) | 1 (1)
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1)
BASEDOW'S DISEASE (Endocrine disorders) | 1 (1)
HYPOTHYROIDISM (Endocrine disorders) | 1 (1)
ADVERSE EVENT (General disorders) | 2 (4)
AUTOIMMUNE HEPATITIS (Hepatobiliary disorders) | 1 (1)
APPENDICITIS (Infections and infestations) | 1 (1)
OSTEOMYELITIS (Infections and infestations) | 1 (1)
TOXOPLASMOSIS (Infections and infestations) | 1 (1)
NARCOTIC INTOXICATION (Injury, poisoning and procedural complications) | 1 (1)
WEIGHT DECREASED (Investigations) | 1 (1)
CONVULSION (Nervous system disorders) | 1 (1)
DISTURBANCE IN ATTENTION (Nervous system disorders) | 1 (1)
AGGRESSION (Psychiatric disorders) | 1 (1)
ALCOHOL ABUSE (Psychiatric disorders) | 1 (2)
ALCOHOL PROBLEM (Psychiatric disorders) | 1 (1)
ANXIETY DISORDER (Psychiatric disorders) | 1 (1)
DEPRESSION (Psychiatric disorders) | 5 (7)
MERYCISM (Psychiatric disorders) | 1 (1)
PSYCHIATRIC DECOMPENSATION (Psychiatric disorders) | 2 (2)
PSYCHOTIC DISORDER (Psychiatric disorders) | 3 (3)
RESTLESSNESS (Psychiatric disorders) | 1 (1)
SUICIDAL IDEATION (Psychiatric disorders) | 1 (1)
SUICIDE ATTEMPT (Psychiatric disorders) | 1 (3)
ALOPECIA (Skin and subcutaneous tissue disorders) | 2 (2)
DRY SKIN (Skin and subcutaneous tissue disorders) | 1 (3)
PRURITUS (Skin and subcutaneous tissue disorders) | 3 (3)
SKIN BURNING SENSATION (Skin and subcutaneous tissue disorders) | 1 (1)
APPENDICECTOMY (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=746)
ANAEMIA (Blood and lymphatic system disorders) | 46 (50)
DIARRHOEA (Gastrointestinal disorders) | 40 (42)
NAUSEA (Gastrointestinal disorders) | 74 (80)
FATIGUE (General disorders) | 105 (131)
IRRITABILITY (General disorders) | 47 (47)
PYREXIA (General disorders) | 44 (49)
INFLUENZA (Infections and infestations) | 68 (71)
WEIGHT DECREASED (Investigations) | 69 (77)
ANOREXIA (Metabolism and nutrition disorders) | 68 (71)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 55 (56)
MYALGIA (Musculoskeletal and connective tissue disorders) | 42 (42)
DISTURBANCE IN ATTENTION (Nervous system disorders) | 51 (53)
DIZZINESS (Nervous system disorders) | 41 (41)
HEADACHE (Nervous system disorders) | 86 (87)
DEPRESSED MOOD (Psychiatric disorders) | 41 (44)
DEPRESSION (Psychiatric disorders) | 52 (58)
SLEEP DISORDER (Psychiatric disorders) | 76 (79)
COUGH (Respiratory, thoracic and mediastinal disorders) | 38 (40)
ALOPECIA (Skin and subcutaneous tissue disorders) | 63 (70)
PRURITUS (Skin and subcutaneous tissue disorders) | 59 (59)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No